CLINICAL TRIAL: NCT02634619
Title: A Randomized Study of Dorsal Versus Ventral Buccal Mucosa Graft Onlay for Bulbar Urethroplasty
Brief Title: A Study of Dorsal Versus Ventral Buccal Mucosa Graft Onlay for Bulbar Urethroplasty
Acronym: DvV
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patient enrollment was slow and we were not able to accrue participants at a decent pace.
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Minnesota (Other); Baylor College of Medicine (Other); University of Iowa (Other); University of Kansas (Other); Central Ohio Urology Group (Other); Loyola University Chicago (Other); Lahey Clinic (Other); University of Washington (Other); New York University (Other); University of California, San Diego (Other); University of Utah (Other)
Responsible Party: Principal Investigator, Benjamin Breyer, MD, Chief of Urology, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K12DK083021-DvV; K12DK083021 (NIH)
Record Dates: First submitted 2015-11-17; First posted 2015-12-18 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Urethral Stricture
Keywords: urethral stricture
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ventral Buccal Mucosa Graft Onlay (Active Comparator): Standard of care method for repairing urethral strictures
  Interventions: Procedure: Ventral buccal mucosa onlay urethroplasty
- Dorsal Buccal Mucosa Graft Onlay (Active Comparator): Standard of care method for repairing urethral strictures
  Interventions: Procedure: Dorsal buccal mucosa onlay urethroplasty

INTERVENTIONS:
Procedure: Ventral buccal mucosa onlay urethroplasty — Ventral buccal graft onlay involves a midline perineal incision and retraction of the bulbospongiosum muscle downward to expose the ventral urethral surface. The corpus spongiosum is incised longitudinally to expose the urethral lumen and the incision is extended proximal and distal to the established stricture. The buccal mucosa graft is harvested and trimmed to the length and width of the urethrotomy and the graft is sutured at the proximal and distal apices and a running suture at the lateral margins to establish a tight anastomosis. Ventral placement allows for limited urethral mobilization and easy access, but there is concern about higher likelihood of diverticulum formation and development of other associated complications - such as post void dribbling and ejaculatory dysfunction.
  Arms: Ventral Buccal Mucosa Graft Onlay
Procedure: Dorsal buccal mucosa onlay urethroplasty — Dorsal buccal onlay also involves a midline perineal incision. The bulbo-cavernosum and corpora cavernosum are dissected from the bulbar urethra allowing for complete mobilization of the urethra. The urethra is rotated 180 degrees to allow for dorsal access and an incision is made on the dorsal urethra proximal and distal to the stricture location. The buccal graft is harvested and trimmed to the appropriate size of the urethrotomy and spread on the overlying tunica albuginea of the corporal bodies. The urethra is rotated back to allow for suturing of the left mucosal margin to the left margin of the buccal graft and corporal bodies, essentially covering the entire urethral plate. Dorsal placement has potential for a more stable vascular bed for graft sustainability and less spongiosal bleeding, but requires a greater urethral mobilization and longer operative times.
  Arms: Dorsal Buccal Mucosa Graft Onlay

SUMMARY:
The investigators propose a randomized non-blinded comparison of dorsal vs. ventral approach for buccal mucosa graft urethroplasty in the bulbar urethra. Buccal mucosa graft is a common method of repairing the strictured urethra. Current evidence suggests the two approaches for placement of the graft are equally successful at correcting the stricture and the two approaches have similar risks of complications. The investigators propose to randomly assign appropriately selected patients to either a dorsally- or ventrally-placed graft. No additional procedures beyond normal care protocol will be required of the patients. Success will be assessed via objective and subjective methods; complications will be tallied in a standardized fashion. Outcomes will be measured at two years.

DETAILED DESCRIPTION:
1. Screening for eligibility; Enrollment/baseline: Patients are referred to UCSF urology clinic for urethroplasty. Participants commonly come to the clinic having already had imaging of their stricture, completed the appropriate PROMs, uroflowmetry and post-void residual urine volume measurement. The patient usually leaves the initial clinic visit with a scheduled surgery. Thus, both screening and enrollment will be done at the initial clinic visit. If the patient agrees to enroll and signs the consent form, they will then be randomized.
2. Randomization: The PI will contact the research assistant by email or telephone and communicate the random identification number of the subject and receive the random assignment to ventral or dorsal graft. This will usually occur after the initial clinic visit but certainly before the surgery date. Patients will not be blinded as to their assignment. Surgeons, out of necessity, will not be blinded as well.
3. Treatment/intervention period: Patient will undergo urethroplasty using standard approach and graft will be placed ventrally or dorsally, as assigned. Most patients go home the same day after surgery. A catheter will be left in the urethra for 2-4 weeks as is standard approach for buccal graft urethroplasties.
4. Follow-up (there will be no extra clinic visits, questionnaires, or tests beyond that which the investigators normally do for all patients undergoing urethroplasty):

   1. 2-4 weeks: urethral catheter removal and urethrogram to document well-healed suture line
   2. 3 and 12 months post-operative clinic visit:

   i. cystoscopy ii. PROMs and additional post-operative questionnaires iii. Uroflowmetry and post-void residual urine volume c. Annual visits after year 1: The investigators will typically follow patients annually with no end date after urethroplasty. For publication purposesits has been set to 1 year as the study end date but the investigators will continue to see the patients outside the study protocol after year 1 (so that participants receive the same care as people not in the study) and will perform the following: i. Cystoscopy, if indicated based on abnormalities in ii or iii ii. PROMs and additional post-operative questionnaires iii. Uroflowmetry and post-void residual urine volume
5. Data Safety and Monitoring Both ventral and dorsal buccal mucosa graft are standard of care and all surgeons in this study have performed at least 50-100 of each of these surgeries. Investigators do not anticipate adverse events that are not well known in the literature. Urethroplasty is generally a low risk surgery. Still, any AEs will be monitored by the surgeon and communicated to Dr. Jeremy Myers at The University of Utah, which serves as the coordinating center for this study.

ELIGIBILITY:
Inclusion Criteria:

* Male ≥ 18 years old with diagnosis of bulbar urethral stricture by voiding cystourethrogram of known and/or idiopathic etiology.
* Male patients with bulbar urethral stricture > 1 cm in length
* Strictures must predominantly include the proximal and/or mid-bulbar urethra
* Strictures may extend from the mid-bulbar urethra into the distal bulbar urethra

Exclusion Criteria:

* Patients with prior history of open urethral surgery, such as:

  * Prior urethroplasty
  * Artificial urniary Sphincter placement
  * Male urethral sling placement
  * Rectourethral fistula
* Radiation therapy to the abdomen or pelvis
* Patients with previous hypospadias repair
* lichen sclerosis
* no involvement of the pendulous urethra

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Anatomic recurrence of urethral stricture observed by cystoscopy or RUG/VCUG | Through study completion, an average of up to 1 year
  This is defined by the patient as slowing of urinary stream in conjunction with stricture recurrence

SECONDARY OUTCOMES:
Outcome of perioperative complication deep vein thrombosis (DVT), determined by medical history, physical examination, and/or ultrasound: | Through study completion, an average of up to 1 year
  DVT occurs when a blood clot forms in one or more of the deep veins in your body, typically in the legs, and carries with it significant morbidity. Determination is based on medical history (overall health, medications, recent surgery, etc.), physical examination for signs of DVT, and if needed, diagnostic tests such as ultrasound.
Outcome of perioperative complication: positioning complaints | Through study completion, an average of up to 1 year
  In order to do the operation, patients are placed in an exaggerated lithotomy position that may cause nerve injury or muscle soreness
Outcome of perioperative complication perineal abscess, determined through physical or digital examination: | Through study completion, an average of up to 1 year
  Perineal abscess is an infectious complication that develops after bacteria overgown and form a collection of pus. Often this will require surgical drainage
Leak at 2-3 week post-op voiding cystourethrogram (VCUG) to identify if there is any leak at the site of repair | Observed at 2-3 weeks post-op
  After 2-3 weeks, patients will return to have their Foley catheters removed. At this time, we will perform a voiding cystourethrogram (vcug) to identify if there is any leak at the site of repair. We can see this leak by injecting contrast dye.
Max urinary flow rate (mL/sec) | Observed at 3 month post-op & 12 month post-op
  Maximal milliliters per seconds that the patient can urinate
Intervention rate: catheter self dilation / dilation | Through study completion, an average of up to 1 year
  Patients will occasionally perform self dilation with a catheter to keep their stricture patent after surgery.
Intervention rate: DVIU | Through study completion, an average of up to 1 year
  Stricture recurrence that causes severe restriction in urinary flow may require a direct visual internal urethrotomy (DVIU) following urethroplasty. DVIU is the repair of a narrow segment (stricture) of the urethra. A small scope is placed into the urethra, and a cut is made to repair the stricture.
Intervention rate: repeat urethroplasty | Through study completion, an average of up to 1 year
  Stricture recurrence that causes severe restriction in urinary flow may require a repeat urethroplasty

OTHER OUTCOMES:
Delta Sexual Health Inventory for Men (SHIM) to determinate erectile dysfunction | Administered at 3 &12 month post op
  This is a validated abridged and slightly modified 5-item version of the 15-item International Index of Erectile Function, designed for easy use, by clinicians, to diagnose the presence and severity of ED in clinical settings
Delta Male Sexual Health Questionnaire (MSHQ) to assess sexual function | Administered at 3 & 12 month post op
  This is a validated questionaire that includes domains for erectile function, ejaculatory function, sexual satisfaction, and provides a more in depth assessment of ejaculatory function and sexual satisfaction than the IIEF.

CONTACTS AND LOCATIONS:
Overall Officials: benjamin n breyer, MD, MAS, FAC, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Andrich DE, Leach CJ, Mundy AR. The Barbagli procedure gives the best results for patch urethroplasty of the bulbar urethra. BJU Int. 2001 Sep;88(4):385-9. doi: 10.1046/j.1464-410x.2001.02344.x. PMID 11564027
- [Background] Andrich DE, Mundy AR. Substitution urethroplasty with buccal mucosal-free grafts. J Urol. 2001 Apr;165(4):1131-3; discussion 1133-4. PMID 11257653
- [Background] Barbagli G, De Stefani S, Sighinolfi MC, Annino F, Micali S, Bianchi G. Bulbar urethroplasty with dorsal onlay buccal mucosal graft and fibrin glue. Eur Urol. 2006 Sep;50(3):467-74. doi: 10.1016/j.eururo.2006.05.018. Epub 2006 Jun 5. PMID 16806665
- [Background] Barbagli G, Palminteri E, Guazzoni G, Montorsi F, Turini D, Lazzeri M. Bulbar urethroplasty using buccal mucosa grafts placed on the ventral, dorsal or lateral surface of the urethra: are results affected by the surgical technique? J Urol. 2005 Sep;174(3):955-7; discussion 957-8. doi: 10.1097/01.ju.0000169422.46721.d7. PMID 16094007
- [Background] Barbagli G, Palminteri E, Rizzo M. Dorsal onlay graft urethroplasty using penile skin or buccal mucosa in adult bulbourethral strictures. J Urol. 1998 Oct;160(4):1307-9. PMID 9751341
- [Background] Dubey D, Kumar A, Bansal P, Srivastava A, Kapoor R, Mandhani A, Bhandari M. Substitution urethroplasty for anterior urethral strictures: a critical appraisal of various techniques. BJU Int. 2003 Feb;91(3):215-8. doi: 10.1046/j.1464-410x.2003.03064.x. PMID 12581007
- [Background] Dubey D, Kumar A, Mandhani A, Srivastava A, Kapoor R, Bhandari M. Buccal mucosal urethroplasty: a versatile technique for all urethral segments. BJU Int. 2005 Mar;95(4):625-9. doi: 10.1111/j.1464-410X.2005.05352.x. PMID 15705092
- [Background] Elliott SP, Metro MJ, McAninch JW. Long-term followup of the ventrally placed buccal mucosa onlay graft in bulbar urethral reconstruction. J Urol. 2003 May;169(5):1754-7. doi: 10.1097/01.ju.0000057800.61876.9b. PMID 12686826
- [Background] Fichtner J, Filipas D, Fisch M, Hohenfellner R, Thuroff JW. Long-term outcome of ventral buccal mucosa onlay graft urethroplasty for urethral stricture repair. Urology. 2004 Oct;64(4):648-50. doi: 10.1016/j.urology.2004.05.011. PMID 15491691
- [Background] Heinke T, Gerharz EW, Bonfig R, Riedmiller H. Ventral onlay urethroplasty using buccal mucosa for complex stricture repair. Urology. 2003 May;61(5):1004-7. doi: 10.1016/s0090-4295(02)02523-2. PMID 12736024
- [Background] Kane CJ, Tarman GJ, Summerton DJ, Buchmann CE, Ward JF, O'Reilly KJ, Ruiz H, Thrasher JB, Zorn B, Smith C, Morey AF. Multi-institutional experience with buccal mucosa onlay urethroplasty for bulbar urethral reconstruction. J Urol. 2002 Mar;167(3):1314-7. PMID 11832721
- [Background] Kellner DS, Fracchia JA, Armenakas NA. Ventral onlay buccal mucosal grafts for anterior urethral strictures: long-term followup. J Urol. 2004 Feb;171(2 Pt 1):726-9. doi: 10.1097/01.ju.0000103500.21743.89. PMID 14713797
- [Background] Mangera A, Patterson JM, Chapple CR. A systematic review of graft augmentation urethroplasty techniques for the treatment of anterior urethral strictures. Eur Urol. 2011 May;59(5):797-814. doi: 10.1016/j.eururo.2011.02.010. Epub 2011 Feb 24. PMID 21353379
- [Background] Morey AF, McAninch JW. When and how to use buccal mucosal grafts in adult bulbar urethroplasty. Urology. 1996 Aug;48(2):194-8. doi: 10.1016/S0090-4295(96)00154-9. PMID 8753728
- [Background] Pansadoro V, Emiliozzi P, Gaffi M, Scarpone P, DePaula F, Pizzo M. Buccal mucosa urethroplasty in the treatment of bulbar urethral strictures. Urology. 2003 May;61(5):1008-10. doi: 10.1016/s0090-4295(02)02585-2. PMID 12736025
- [Background] Raber M, Naspro R, Scapaticci E, Salonia A, Scattoni V, Mazzoccoli B, Guazzoni G, Rigatti P, Montorsi F. Dorsal onlay graft urethroplasty using penile skin or buccal mucosa for repair of bulbar urethral stricture: results of a prospective single center study. Eur Urol. 2005 Dec;48(6):1013-7. doi: 10.1016/j.eururo.2005.05.003. Epub 2005 May 31. PMID 15970374
- [Background] Wang K, Miao X, Wang L, Li H. Dorsal onlay versus ventral onlay urethroplasty for anterior urethral stricture: a meta-analysis. Urol Int. 2009;83(3):342-8. doi: 10.1159/000241680. Epub 2009 Oct 13. PMID 19829038
- [Background] Wessells H, McAninch JW. Use of free grafts in urethral stricture reconstruction. J Urol. 1996 Jun;155(6):1912-5. PMID 8618286
- [Background] Xu YM, Qiao Y, Sa YL, Wu DL, Zhang XR, Zhang J, Gu BJ, Jin SB. Substitution urethroplasty of complex and long-segment urethral strictures: a rationale for procedure selection. Eur Urol. 2007 Apr;51(4):1093-8; discussion 1098-9. doi: 10.1016/j.eururo.2006.11.039. Epub 2006 Nov 27. PMID 17157433